CLINICAL TRIAL: NCT02431702
Title: A Prospective, Matched-Control, Randomized, Open-Label, Flexible-Dose, Study in Subjects With Recent-Onset Schizophrenia or Schizophreniform Disorder to Compare Disease Progression and Disease Modification Following Treatment With Paliperidone Palmitate Long-Acting Injection or Oral Antipsychotics
Brief Title: A Study to Compare Disease Progression and Modification Following Treatment With Paliperidone Palmitate Long-Acting Injection or Oral Antipsychotics in Participant's With Recent-onset Schizophrenia or Schizophreniform
Acronym: DREaM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR106193; R092670SCH3013 (Other: Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2015-04-28; First posted 2015-05-01 (Estimated); Results first posted 2021-01-19 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Schizophrenia; Psychotic Disorders
Keywords: Paliperidone Palmitate; Oral Antipsychotics; Schizophrenia; Psychotic Disorders; Cognition in Schizophrenia; Brain intracortical myelin volume; Personal and Social Performance; Disease Modification
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Aripiprazole; Haloperidol; Olanzapine; Paliperidone Palmitate; Perphenazine; Quetiapine Fumarate; Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (6):
- Part-1: Oral Antipsychotics (OAP) (Active Comparator): All Participants will receive Paliperidone Extended Release (ER) 1.5 to 12 milligram (mg) or risperidone 1 to 6 mg once daily orally for 2 months. Subjects who tolerate paliperidone ER/risperidone but find it inadequately efficacious after treatment for an adequate duration at an adequate dosage (per clinical judgment), may be switched to another protocol-specified OAP at the discretion of the investigator.
  Interventions: Drug: Aripiprazole; Drug: Haloperidol; Drug: Olanzapine; Drug: Oral Paliperidone ER; Drug: Perphenazine; Drug: Quetiapine; Drug: Oral Risperidone
- Part-2: Paliperidone Palmitate (PP) (Experimental): Participants who will complete Part-1 will be randomized to receive oral Paliperidone Palmitate (PP) treatment. Participants will receive 5 doses of PP1M (paliperidone palmitate once-monthly injection). First dose at a starting dose of 234 mg on Day 1 and thereafter second dose in second week and then, every month up to Day 92. Participants will be subsequently switched to PP3M (paliperidone palmitate three-monthly injection) following a minimum of 5 injections of PP1M. Participants receiving PP3M may go back to treatment with PP1M (monthly injections of 78, 117, 156 or 234 mg, flexibly dosed) for further dose adjustment or for the duration of the study with the approval of the medical monitor.
  Interventions: Drug: Paliperidone Palmitate Injection (PP1M); Drug: Paliperidone Palmitate Injection (PP3M)
- Part-2: OAP (Active Comparator): Participants who will complete Part-1 will be randomized to receive Oral Antipsychotics for 9 months.
  Interventions: Drug: Aripiprazole; Drug: Haloperidol; Drug: Olanzapine; Drug: Oral Paliperidone ER; Drug: Perphenazine; Drug: Quetiapine; Drug: Oral Risperidone
- Part-3: PP - PP (Experimental): Participants who will complete Part-2 (with PP treatment) will continue to receive Paliperidone Palmitate for 9 months.
  Interventions: Drug: Paliperidone Palmitate Injection (PP3M)
- Part-3: OAP - Delayed Start Paliperidone Palmitate (PP) (Experimental): Participants who will complete Part-2 (with OAP treatment) will be randomized to receive PP treatment for 9 months. PP treatment includes PP1M and PP3M. Participants will be subsequently switched to PP3M following a minimum of 5 injections of PP1M. Participants receiving PP3M may go back to treatment with PP1M (monthly injections of 78, 117, 156 or 234 mg, flexibly dosed) for further dose adjustment or for the duration of the study with the approval of the medical monitor.
  Interventions: Drug: Paliperidone Palmitate Injection (PP1M); Drug: Paliperidone Palmitate Injection (PP3M)
- Part-3: OAP - OAP (Active Comparator): Participants who will complete Part-2 (with OAP treatment) will be randomized to receive OAP treatment for additional 9 months.
  Interventions: Drug: Aripiprazole; Drug: Haloperidol; Drug: Olanzapine; Drug: Oral Paliperidone ER; Drug: Perphenazine; Drug: Quetiapine; Drug: Oral Risperidone

INTERVENTIONS:
Drug: Aripiprazole — Aripiprazole will be administered in accordance with the label or Investigator's discretion
  Arms: Part-1: Oral Antipsychotics (OAP); Part-2: OAP; Part-3: OAP - OAP
Drug: Haloperidol — Haloperidol will be administered in accordance with the label or Investigator's discretion
  Arms: Part-1: Oral Antipsychotics (OAP); Part-2: OAP; Part-3: OAP - OAP
Drug: Olanzapine — Olanzapine will be administered in accordance with the label or Investigator's discretion
  Arms: Part-1: Oral Antipsychotics (OAP); Part-2: OAP; Part-3: OAP - OAP
Drug: Oral Paliperidone ER — Paliperidone Extended Release (ER) tablets 1.5 to 12 milligram (mg) per day will be administered orally.
  Arms: Part-1: Oral Antipsychotics (OAP); Part-2: OAP; Part-3: OAP - OAP
Drug: Perphenazine — Perphenazine will be administered in accordance with the label or Investigator's discretion
  Arms: Part-1: Oral Antipsychotics (OAP); Part-2: OAP; Part-3: OAP - OAP
Drug: Quetiapine — Quetiapine will be administered in accordance with the label or Investigator's discretion
  Arms: Part-1: Oral Antipsychotics (OAP); Part-2: OAP; Part-3: OAP - OAP
Drug: Oral Risperidone — Risperidone tablets 1-6 mg per day will be administered orally.
  Arms: Part-1: Oral Antipsychotics (OAP); Part-2: OAP; Part-3: OAP - OAP
Drug: Paliperidone Palmitate Injection (PP1M) — Participants will receive 5 doses of PP1M. First dose at a starting dose of 234 mg on Day 1 and a second dose of 156 mg on Day 8 and then 78 to 234 mg (in 3 flexible doses), every month up to Day 92.
  Arms: Part-2: Paliperidone Palmitate (PP); Part-3: OAP - Delayed Start Paliperidone Palmitate (PP)
Drug: Paliperidone Palmitate Injection (PP3M) — Paliperidone Palmitate injection (PP3M) will be administered once every 12 weeks intramuscularly. The initial dose will be calculated as 3.5 fold multiple of the final PP1M dose administered on Day 92 (or Day 176). Dose will be increased based on Investigator's discretion.
  Arms: Part-2: Paliperidone Palmitate (PP); Part-3: OAP - Delayed Start Paliperidone Palmitate (PP); Part-3: PP - PP

SUMMARY:
The purpose of the study is to compare effectiveness of paliperidone palmitate (PP: paliperidone palmitate once-monthly and 3-month injections) versus oral antipsychotic (OAP [that is oral paliperidone extended release {ER}, oral risperidone, or another OAP]) in delaying time to treatment failure. The study will also evaluate changes in cognition, functioning, brain intracortical myelin (ICM) volume following treatment with PP compared with OAP in participants with recent-onset schizophrenia or schizophreniform disorder.

DETAILED DESCRIPTION:
A Prospective, matched-control, Randomized (assignment of study drug by chance), open-label, flexible-dose, study in participants with recent-onset schizophrenia or schizophreniform disorder to compare disease progression and disease modification following treatment with PP long-acting injection (once-monthly followed by 3-month injections) or OAP (Any of the following 7 OAPs are permitted: aripiprazole, haloperidol, olanzapine, paliperidone ER, perphenazine, quetiapine, and risperidone). The study consists of 3 parts. Part-1 (Oral Run-In Phase), Part-2 (Disease Progression) and Part-3 (Extended Disease Progression and Disease Modification) with unique endpoints. Screening period will be up to 4 Weeks. Duration of Parts will be as: 2 months for Part-1, 9 months for Part-2 and Part-3. All participants will initially receive oral paliperidone ER or oral risperidone in Part-1. After paliperidone/risperidone treatment in Part-1, participants will be randomized into 1:2 ratio to receive PP or OAP in Part-2. Participants who complete Part-2 will enter into Part-3 wherein OAP group participants of Part-2 will be re-randomized into 1:1 ratio to OAP-OAP group and OAP-PP group, and PP group will continue without further randomization. Treatment failures will be evaluated in Part-2 and Part-3 of the study. Also changes in cognition, functioning, brain intracortical myelin (ICM) volume will be evaluated in the study. Participants' safety will be monitored throughout. Healthy controls (comparable in age, sex, race, and highest parental education to the treated participants) were recruited at each of the 3 MRI centers as controls for the MRI machine calibration for the duration of the study. These healthy controls were to undergo MRI assessments, but were not otherwise involved with the study and did not receive study medication. No safety or efficacy data were collected for these healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a current diagnosis of schizophrenia (295.90) or schizophreniform disorder (295.40) as defined by Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) and confirmed by the Structured Clinical Interview for DSM-5 Disorders (SCID) with a first psychotic episode within the last 24 months prior to the screening visit
* Participant requires treatment with an antipsychotic medication
* Participant must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and are willing to participate in the study
* Participant must have available a designated individual (example, family member, significant other, friend) who has knowledge of the participant and is generally aware of the participants daily activities, and who agrees to let the study site personnel know of changes in the participants circumstances when the participant is not able to provide this information. The designated individual must sign an informed consent form
* Participant is anticipated to have a stable place of residence for the duration of the trial

Exclusion Criteria:

* Participant has a current DSM-5 diagnosis of dissociative disorder, bipolar disorder, major depressive disorder, schizoaffective disorder, autistic disorder, or intellectual disabilities
* Participant meets the DSM-5 definition of moderate or severe substance use disorder (except for nicotine) within 2 months prior to Screening
* Participant has a history of neuroleptic malignant syndrome
* Participant has received long-acting injectable (LAI) medication within 2 injection cycles prior to the Screening visit
* Participant has mental retardation, defined as pre-morbid intelligence quotient (IQ) as measured by Wechsler Test of Adult Reading at Screening less than (<) 70

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 337 (Actual)
Dates: Start 2015-07-08 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (38):
- United States (34):
  - Little Rock, Arkansas
  - Garden Grove, California
  - Lemon Grove, California
  - Los Angeles, California
  - San Diego, California
  - San Rafael, California
  - Stanford, California
  - Lauderdale Lakes, Florida
  - Leesburg, Florida
  - Miami, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Chicago, Illinois
  - Granite City, Illinois
  - Hoffman Estates, Illinois
  - Indianapolis, Indiana
  - Louisville, Kentucky
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - East Lansing, Michigan
  - Grand Rapids, Michigan
  - Muskegon, Michigan
  - Omaha, Nebraska
  - Albuquerque, New Mexico
  - Cedarhurst, New York
  - Rochester, New York
  - Staten Island, New York
  - Charlotte, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Eugene, Oregon
  - Philadelphia, Pennsylvania
  - Houston, Texas
  - Bothell, Washington
- Brazil (3):
  - Itapira
  - Rio de Janeiro
  - São José
- México, Mexico

REFERENCES:
- [Derived] Lopena OJ, Alphs LD, Sajatovic M, Turkoz I, Sun L, Johnston KL, Sliwa JK, Najarian DM, Starr HL. Earlier Use of Long-Acting Injectable Paliperidone Palmitate Versus Oral Antipsychotics in Patients With Schizophrenia: An Integrated Patient-Level Post Hoc Analysis. J Clin Psychiatry. 2023 Sep 25;84(6):23m14788. doi: 10.4088/JCP.23m14788. PMID 37756123
- [Derived] Tishler TA, Ellingson BM, Salvadore G, Baker P, Turkoz I, Subotnik KL, de la Fuente-Sandoval C, Nuechterlein KH, Alphs L. Effect of treatment with paliperidone palmitate versus oral antipsychotics on frontal lobe intracortical myelin volume in participants with recent-onset schizophrenia: Magnetic resonance imaging results from the DREaM study. Schizophr Res. 2023 May;255:195-202. doi: 10.1016/j.schres.2023.03.023. Epub 2023 Mar 31. PMID 37004331
- [Derived] Alphs L, Baker P, Brown B, Fu DJ, Turkoz I, Nuechterlein KH. Evaluation of major treatment failure in patients with recent-onset schizophrenia or schizophreniform disorder: A post hoc analysis from the Disease Recovery Evaluation and Modification (DREaM) study. Schizophr Res. 2022 Oct;248:58-63. doi: 10.1016/j.schres.2022.07.015. Epub 2022 Aug 6. PMID 35939921
- [Derived] Alphs L, Brown B, Turkoz I, Baker P, Fu DJ, Nuechterlein KH. The Disease Recovery Evaluation and Modification (DREaM) study: Effectiveness of paliperidone palmitate versus oral antipsychotics in patients with recent-onset schizophrenia or schizophreniform disorder. Schizophr Res. 2022 May;243:86-97. doi: 10.1016/j.schres.2022.02.019. Epub 2022 Mar 2. PMID 35247794

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 337 participants were enrolled out of which 273 were randomized and received study medication while 64 did not and served as healthy controls. Healthy controls underwent MRI assessments as controls for the MRI machine calibration. They did not receive study medication and no safety or efficacy data were collected.
Pre-assignment Details: To ensure that the total number of participants equal 337, another group is created called "Healthy Controls" to the table below and their completion status is reported in Part 1 and not in other parts.
Groups:
- Part 1-Run-in: Oral Antipsychotics (OAP): All participants received paliperidone extended Release (ER) 1.5 to 12 milligrams (mg) or risperidone 1 to 6 mg once daily orally for 2 months. Participants who tolerated paliperidone ER/risperidone but found it inadequately efficacious after treatment for an adequate duration at an adequate dosage (per clinical judgment), may be switched to another protocol-specified OAP at the discretion of the investigator.
- Part 2-Paliperidone Palmitate (PP): Participants who completed Part 1 with acceptable run-in dosages were eligible to enter Part 2. Participants who were randomized to the PP treatment group received a minimum of 5 doses of PP1M with fixed initial doses of 234 mg on Day 1 and 156 mg on Day 8, followed by 3 injections of flexible doses. On Day 120, participants received PP3M for the remaining 9 months.
- Part 2-OAP: Participants who completed Part 1 with acceptable run-in dosages were eligible to enter Part 2. Participants who completed Part 1 were randomized to OAP treatment group and continued their OAP treatment from Part 1 for another 9 months (up to Day 260 of Part 2).
- Part 3-PP to PP (Extended Disease Progression [EDP] and Disease Modification): Participants who completed Part 2 and who were eligible based on matched criteria identified in Part 1 continued on the PP Treatment Group in Part 3. Participants continued to receive Paliperidone Palmitate for another 9 months (up to Day 260 Part 3).
- Part 3- OAP to PP (or Delayed-Start PP) (Disease Modification): Participants who completed Part 2 (with OAP treatment) and who were eligible based on matched criteria identified in Part 1 were re-randomized to receive PP treatment for additional 9 months (up to Day 260). PP treatment includes PP1M or PP3M. Participants subsequently switched to PP3M following a minimum of 5 injections of PP1M.
- Part 3-OAP to OAP (EDP and Disease Modification): Participants who completed Part 2 (with OAP treatment) and who were eligible based on matched criteria identified in Part 1 were re-randomized to receive OAP treatment for another 9 months (up to Day 260 of Part 3).
- Healthy Controls: Participants did not receive any study medication and did not fall into any of the 3 parts of the study. For reporting purposes, the completion of the Healthy Controls were entered in Part 1 and not in the other parts.
Period: Part 1: 2-Month Oral Run-in Phase
Arm/Group | Part 1-Run-in: Oral Antipsychotics (OAP) | Part 2-Paliperidone Palmitate (PP) | Part 2-OAP | Part 3-PP to PP (Extended Disease Progression [EDP] and Disease Modification) | Part 3- OAP to PP (or Delayed-Start PP) (Disease Modification) | Part 3-OAP to OAP (EDP and Disease Modification) | Healthy Controls
Started | 273 | 0 | 0 | 0 | 0 | 0 | 64
Completed | 239 | 0 | 0 | 0 | 0 | 0 | 32
Not Completed | 34 | 0 | 0 | 0 | 0 | 0 | 32
Not completed — Adverse Event | 7 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 11 | 0 | 0 | 0 | 0 | 0 | 23
Not completed — Withdrawal of Consent | 9 | 0 | 0 | 0 | 0 | 0 | 6
Not completed — Other | 5 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Does not Tolerate Paliperidone ER | 2 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: 9Month Disease Progression Phase
Arm/Group | Part 1-Run-in: Oral Antipsychotics (OAP) | Part 2-Paliperidone Palmitate (PP) | Part 2-OAP | Part 3-PP to PP (Extended Disease Progression [EDP] and Disease Modification) | Part 3- OAP to PP (or Delayed-Start PP) (Disease Modification) | Part 3-OAP to OAP (EDP and Disease Modification) | Healthy Controls
Started | 0 | 78 (Participants who completed Part 1 and were eligible to be randomized in this group.) | 157 (Participants who completed Part 1 and were eligible to be randomized in this group.) | 0 | 0 | 0 | 0
Completed | 0 | 52 | 128 | 0 | 0 | 0 | 0
Not Completed | 0 | 26 | 29 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 5 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 6 | 13 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 11 | 8 | 0 | 0 | 0 | 0
Not completed — Assigned PP, but required OAP | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 2 | 2 | 0 | 0 | 0 | 0
Not completed — Assigned OAP, but required PP | 0 | 0 | 5 | 0 | 0 | 0 | 0
Period: Part 3: 9 Month of Additional Treatment
Arm/Group | Part 1-Run-in: Oral Antipsychotics (OAP) | Part 2-Paliperidone Palmitate (PP) | Part 2-OAP | Part 3-PP to PP (Extended Disease Progression [EDP] and Disease Modification) | Part 3- OAP to PP (or Delayed-Start PP) (Disease Modification) | Part 3-OAP to OAP (EDP and Disease Modification) | Healthy Controls
Started | 0 | 0 | 0 | 49 (Participants who completed Part 2 and were eligible to continue treatment in this group.) | 57 (Participants who completed Part 2 and were eligible to be re-randomized in this group.) | 63 (Participants who completed Part 2 and were eligible to be re-randomized in this group.) | 0
Completed | 0 | 0 | 0 | 40 | 47 | 46 | 0
Not Completed | 0 | 0 | 0 | 9 | 10 | 17 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 3 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 5 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 5 | 6 | 6 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 1 | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1-Oral Antipsychotics (OAP): All participants received paliperidone extended Release (ER) 1.5 to 12 milligrams (mg) or risperidone 1 to 6 mg once daily orally for 2 months. Participants who tolerated paliperidone ER/risperidone but found it inadequately efficacious after treatment for an adequate duration at an adequate dosage (per clinical judgment), may be switched to another protocol-specified OAP at the discretion of the investigator.
Arm/Group | Part 1-Oral Antipsychotics (OAP)
Number analyzed (Participants) | 273
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.2 (4.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 213
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 95
  Not Hispanic or Latino | 173
  Unknown or Not Reported | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 17
  Black or African American | 91
  Native Hawaiian or Other Pacific Islander | 2
  White | 124
  More than one race | 0
  Unknown or Not Reported | 0
  Other | 39
Region of Enrollment [Count of Participants; unit: Participants]
  BRAZIL | 40
  MEXICO | 26
  UNITED STATES | 207

OUTCOME MEASURES:

1. Primary Outcome: Part-2 (Disease Progression): Time to First Treatment Failure
Description: Treatment failure is defined as the time from participant's randomization to first treatment failure, which was a composite endpoint consisting of any of the following: 1) Psychiatric hospitalization due to worsening symptoms; 2) Any deliberate self-injury, suicidal ideation or behavior, homicidal ideation or violent behavior that is clinically significant and needs immediate intervention as determined by the study physician; 3) New arrest/incarceration; 4) Discontinuation of antipsychotic treatment due to inadequate efficacy as determined by the study physician; 5) Discontinuation of antipsychotic treatment due to safety or tolerability as determined by the study physician; 6) Treatment supplementation with another antipsychotic due to inadequate efficacy as determined by the study physician; 7) Increase in the level of psychiatric services in order to prevent imminent psychiatric hospitalization as determined by the study physician.
Time Frame: From Day 1 up to 9 Months
Population: Part 2 Intent-to-Treat (ITT) analysis set included all randomized participants who received at least one dose of study medication (or any portion of the dose) in Part 2, regardless of their compliance with the protocol.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Part-2: Paliperidone Palmitate (PP): Participants who completed part 1 with acceptable run-in dosages were eligible to enter Part 2. Participants who were randomized to the PP treatment group received a minimum of 5 doses of PP1M with fixed initial doses of 234 mg on Day 1 and 156 mg on Day 8, followed by 3 injections of flexible doses. On Day 120, participants received PP3M for the remaining 9 months. Participants were subsequently switched to PP3M (paliperidone palmitate three-monthly injection) following a minimum of 5 injections of PP1M.
- Part-2: OAP: Participants who completed Part 1 with acceptable run-in dosages were eligible to enter Part 2. Participants who completed Part 1 were re-randomized to OAP treatment group and continued their OAP treatment from Part 1 for another 9 months (up to Day 260 of Part 2).
Arm/Group | Part-2: Paliperidone Palmitate (PP) | Part-2: OAP
Number analyzed (Participants) | 78 | 157
days | NA [263.0 to NA] — Here, NA signifies median or upper limit of CI was not estimable due to less than 50% of participants experienced an event.. | NA [NA to NA] — Here, NA signifies that median or upper/lower limit of CI was not estimable due to less than 50% of participants experienced an event.

2. Primary Outcome: Part 3 (Extended Disease Progression [EDP]): Change From Baseline in Cognition as Measured by the MATRICS Consensus Cognitive Battery (MCCB) Composite Score
Description: The MATRICS Consensus Cognitive Battery is an instrument that contains 10 tests to measure cognitive performance in 7 cognitive domains: speed processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition. The composite score combines the individual scores of the 10 tests and scores them on a normative scale to derive a T-score and composites scores. The range of T-scores for a normal control population is between 0 to 100 with a mean of 50 and standard deviation of 10. Higher scores indicate better cognitive functioning.
Time Frame: Baseline and 18 Months
Population: Part 3 ITT analysis set included all randomized participants who received at least one dose of study medication (or any portion of the dose) in Part 3, regardless of their compliance with the protocol. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Error); unit: T-score
Groups:
- Part 3-PP to PP: Participants who completed Part 2 and who were eligible based on matched criteria identified in Part 1 continued on the PP Treatment Group in Part 3. Participants continued to receive Paliperidone Palmitate for another 9 months (up to Day 260 Part 3).
- Part 3-OAP to OAP: Participants who completed Part 2 (with OAP treatment) and who were eligible based on matched criteria identified in Part 1 were re-randomized to receive OAP treatment for another 9 months (up to Day 260 of Part 3).
Arm/Group | Part 3-PP to PP | Part 3-OAP to OAP
Number analyzed (Participants) | 39 | 44
T-score | 1.6 (1.19) | 3.2 (1.11)

3. Primary Outcome: Part 3 (Disease Modification): Change From Baseline in Cognition as Measured by the MATRICS Consensus Cognitive Battery (MCCB) Composite Score
Description: as for outcome 2
Time Frame: Baseline and Day 260
Population: Part 3 ITT analysis set included all randomized participants who received at least one dose of study medication (or any portion of the dose) in Part 3, regardless of their compliance with the protocol.
Measure: Mean (Standard Error); unit: T-score
Groups:
- Part 3- PP to PP: Participants who completed Part 2 and who were eligible based on matched criteria identified in Part 1 continued on the PP Treatment Group in Part 3. Participants continued to receive Paliperidone Palmitate for another 9 months (up to Day 260 Part 3).
- Part 3- OAP to PP (or Delayed-Start PP): Participants who completed Part 2 (with OAP treatment) and who were eligible based on matched criteria identified in Part 1 were re-randomized to receive PP treatment for additional 9 months (up to Day 260). PP treatment includes PP1M and PP3M. Participants subsequently switched to PP3M following a minimum of 5 injections of PP1M.
Arm/Group | Part 3- PP to PP | Part 3- OAP to PP (or Delayed-Start PP) | Part 3-OAP to OAP
Number analyzed (Participants) | 49 | 57 | 63
T-score | -0.7 (1.02) | -0.2 (0.95) | 0.5 (0.96)

4. Secondary Outcome: Part 2 (Disease Progression): Change From Baseline in Cognition as Measured by the MATRICS Consensus Cognitive Battery (MCCB) Composite Score
Description: as for outcome 2
Time Frame: Baseline and Month 9
Population: Analysis was performed on Part 2 ITT analysis set. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Part-2: Paliperidone Palmitate (PP) | Part-2: OAP
Number analyzed (Participants) | 52 | 118
T-score | 2.0 (1.01) | 2.8 (0.73)

5. Secondary Outcome: Part 2 (Disease Progression): Change From Baseline in Functioning as Measured by the Personal and Social Performance (PSP) Total Score
Description: The Personal and Social Performance (PSP) scale assesses degree of a participant's dysfunction within 4 domains of behavior: 1) socially useful activities, 2) personal and social relationships, 3) self-care, and 4) disturbing and aggressive behavior. Each domain was assessed on a 6-point scale, from 1 (absent) to 6 (very severe) (1 = absent, 2 = mild, 3 = manifest, 4 = marked, 5 = severe, and 6 = very severe). PSP total score was calculated as sum of all the domain scores and ranges from 1 to 100. Participants with score of 71 to 100 have mild degree of difficulty; from 31 to 70, varying degrees of disability; less than or equal to 30, functioning so poorly as to require intensive supervision. Higher score indicate better performance.
Time Frame: Baseline and Month 9
Population: as for outcome 4
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Part-2: Paliperidone Palmitate (PP) | Part-2: OAP
Number analyzed (Participants) | 51 | 125
units on a scale | 2.5 (1.60) | 2.9 (1.13)

6. Secondary Outcome: Part 2 (Disease Progression): Change From Baseline in Adjusted Intracortical Myelin (ICM) Fraction Score as Measured by Inversion Recovery (IR) and Spin Echo Magnetic Resonance Imaging (MRI)
Description: The adjusted ICM fraction score is quantified as: 1. The volume of myelinated brain tissue is measured separately on co-localized IR and proton density (PD) MRI images, by outlining the boundary between gray matter and white matter on each image. 2. ICM is calculated from the difference of "IR volume minus PD volume". 3. ICM is then expressed as a fraction of the total intracranial volume (ICM divided by intracranial volume). 4. The ICM fraction is then adjusted for effects of age, gender, and race/ethnicity in the sample of treated participants and healthy controls. A decrease in the adjusted ICM fraction score may be a sign of disease progression.
Time Frame: Baseline and Day 260
Population: Analysis was performed on Part 2 ITT analysis set. Here, N (number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Part-2: Paliperidone Palmitate (PP) | Part-2: OAP
Number analyzed (Participants) | 9 | 25
ratio | -0.001 (0.002) | -0.004 (0.001)

7. Secondary Outcome: Part 2 (Disease Progression): Change From Baseline in Working Memory Score: MCCB Domain
Description: MCCB measures cognitive function across cognitive domains and is comprised of 10 independent tests assessing 7 cognitive domains (speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition). A subset of the MCCB cognitive domain was used to assess working memory of participants. The range of working memory score T-scores for a normal control population is between 0 to 100 with a mean of 50 and standard deviation of 10. Higher scores indicate better cognitive functioning.
Time Frame: Baseline and Day 260
Population: Analysis was performed on Part 2 ITT analysis set.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Part-2: Paliperidone Palmitate (PP) | Part-2: OAP
Number analyzed (Participants) | 78 | 157
T-score | -0.2 (1.08) | -0.8 (0.77)

8. Secondary Outcome: Part 2 (Disease Progression): Change From Baseline in Verbal Learning Score: MCCB Domain
Description: MCCB measures cognitive function across cognitive domains and is comprised of 10 independent tests assessing 7 cognitive domains (speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition). A subset of the MCCB cognitive domain was used to assess verbal learning score of participants. The range of verbal learning score T-scores for a normal control population is between 0 to 100 with a mean of 50 and standard deviation of 10. Higher scores indicate better cognitive functioning.
Time Frame: Baseline and Day 260
Population: Analysis was performed on Part 2 ITT analysis set.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Part-2: Paliperidone Palmitate (PP) | Part-2: OAP
Number analyzed (Participants) | 78 | 157
T-score | 1.3 (1.22) | 1.0 (0.85)

9. Secondary Outcome: Part 2 (Disease Progression): Change From Baseline in Speed of Processing Score: MCCB Domain
Description: MCCB measures cognitive function across cognitive domains and is comprised of 10 independent tests assessing 7 cognitive domains (speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition). A subset of the MCCB cognitive domain was used to assess speed of processing score of participants. The range of speed of processing T-scores for a normal control population is between 0 to 100 with a mean of 50 and standard deviation of 10. Higher scores indicate better cognitive functioning.
Time Frame: Baseline and Day 260
Population: Analysis was performed on Part 2 ITT analysis set.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Part-2: Paliperidone Palmitate (PP) | Part-2: OAP
Number analyzed (Participants) | 78 | 157
T-score | 1.8 (1.21) | 3.5 (0.87)

10. Secondary Outcome: Part 2 (Disease Progression): Change From Baseline in Attention/Vigilance Score: MCCB Domain
Description: MCCB measures cognitive function across cognitive domains and is comprised of 10 independent tests assessing 7 cognitive domains (speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition). A subset of the MCCB cognitive domain was used to assess attention/vigilance score of participants. The range of attention/vigilance score T-scores for a normal control population is between 0 to 100 with a mean of 50 and standard deviation of 10. Higher scores indicate better cognitive functioning.
Time Frame: Baseline and Day 260
Population: Analysis was performed on Part 2 ITT analysis set.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Part-2: Paliperidone Palmitate (PP) | Part-2: OAP
Number analyzed (Participants) | 78 | 157
T-score | 3.2 (1.18) | 0.7 (0.85)

11. Secondary Outcome: Part 2 (Disease Progression): Change From Baseline in Visual Learning Score: MCCB Domain
Description: MCCB measures cognitive function across cognitive domains and is comprised of 10 independent tests assessing 7 cognitive domains (speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition). A subset of the MCCB cognitive domain was used to assess visual learning score of participants. The range of visual learning score T-scores for a normal control population is between 0 to 100 with a mean of 50 and standard deviation of 10. Higher scores indicate better cognitive functioning.
Time Frame: Baseline and Day 260
Population: Analysis was performed on part 2 ITT analysis set.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Part-2: Paliperidone Palmitate (PP) | Part-2: OAP
Number analyzed (Participants) | 78 | 157
T-score | 1.3 (1.29) | 1.4 (0.93)

12. Secondary Outcome: Part 2 (Disease Progression): Change From Baseline in Reasoning and Problem Solving: MCCB Domain
Description: MCCB measures cognitive function across cognitive domains and is comprised of 10 independent tests assessing 7 cognitive domains (speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition). A subset of the MCCB cognitive domain was used to assess reasoning and problem solving of participants. The range of reasoning and problem solving T-scores for a normal control population is between 0 to 100 with a mean of 50 and standard deviation of 10. Higher scores indicate better cognitive functioning.
Time Frame: Baseline and Day 260
Population: Analysis was performed on Part 2 ITT analysis set.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Part-2: Paliperidone Palmitate (PP) | Part-2: OAP
Number analyzed (Participants) | 78 | 157
T-score | 0.2 (1.16) | 2.8 (0.83)

13. Secondary Outcome: Part 2 (Disease Progression): Change From Baseline in Social Cognition Score: MCCB Domain
Description: MCCB measures cognitive function across cognitive domains and is comprised of 10 independent tests assessing 7 cognitive domains (speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition). A subset of the MCCB cognitive domain was used to assess social cognition score of participants. The range of social cognition score T-scores for a normal control population is between 0 to 100 with a mean of 50 and standard deviation of 10. Higher scores indicate better cognitive functioning.
Time Frame: Baseline and Day 260
Population: Analysis was performed on Part 2 ITT analysis set.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Part-2: Paliperidone Palmitate (PP) | Part-2: OAP
Number analyzed (Participants) | 78 | 157
T-score | 0.3 (1.25) | 1.6 (0.89)

14. Secondary Outcome: Part 2 (Disease Progression): Change From Baseline in Clinical Global Impression Severity (CGI-S) Score
Description: The Clinical Global Impression Severity (CGI-S) rating scale is used to rate the severity of a participant's overall clinical condition on a 7 point scale. The score ranges from 1 to 7, where 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill participants". Higher scores indicate worsening.
Time Frame: Baseline, up to 9 Months of Part 2
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part-2: Paliperidone Palmitate (PP) | Part-2: OAP
Number analyzed (Participants) | 52 | 126
units on a scale | -0.2 (1.06) | -0.3 (0.94)

15. Secondary Outcome: Part 2 (Disease Progression): Number of Participants With Change From Baseline in Severity of Psychotic Symptoms, as Measured by Clinician-Rated Dimensions of Psychosis Symptom Severity Scale (CRDPSS)
Description: The CRDPSS is an 8-item measure that assesses the severity of mental health symptoms that are important across psychotic disorders, including delusions, hallucinations, disorganized speech, abnormal psychomotor behavior, negative symptoms. Each item on the measure is rated on a 5-point scale (0=none; 1=equivocal; 2=present, but mild; 3=present and moderate; and 4=present and severe). Total Score is taken as summation. A higher score indicates a more severe condition. Worsened or improved is defined as increase or decrease compared to baseline.
Time Frame: Baseline, up to 9 Months
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Part-2: Paliperidone Palmitate (PP) | Part-2: OAP
Number analyzed (Participants) | 50 | 125
Participants
  Hallucinations: Worsened | 7 | 19
  Hallucinations: Unchanged | 29 | 73
  Hallucinations: Improved | 14 | 33
  Delusions: Worsened | 10 | 20
  Delusions: Unchanged | 23 | 70
  Delusions: Improved | 17 | 35
  Disorganized Speech: Worsened | 2 | 13
  Disorganized Speech: Unchanged | 36 | 85
  Disorganized Speech: Improved | 12 | 27
  Abnormal Psychomotor Behavior: Worsened | 9 | 14
  Abnormal Psychomotor Behavior: Unchanged | 37 | 86
  Abnormal Psychomotor Behavior: Improved | 4 | 25
  Negative Symptoms: Worsened | 17 | 25
  Negative Symptoms: Unchanged | 16 | 61
  Negative Symptoms: Improved | 17 | 39
  Impaired Cognition: Worsened | 13 | 29
  Impaired Cognition: Unchanged | 22 | 52
  Impaired Cognition: Improved | 15 | 44
  Mania: Worsened | 1 | 7
  Mania: Unchanged | 47 | 107
  Mania: Improved | 2 | 11
  Depression: Worsened | 7 | 28
  Depression: Unchanged | 33 | 74
  Depression: Improved | 10 | 23

16. Secondary Outcome: Part 2 (Disease Progression): Change From Baseline in Medication Satisfaction Questionnaire (MSQ) Total Score
Description: The Medication Satisfaction Questionnaire (MSQ) is a 7-point, verbally administered, Likert-type scale rated as follows: 1=Extremely Dissatisfied, 2=Very Dissatisfied, 3=Somewhat Dissatisfied, 4=Neither Satisfied Nor Dissatisfied, 5=Somewhat Satisfied, 6=Very Satisfied, 7=Extremely Satisfied. Worst value is 1 (Extremely Dissatisfied) and best value is 7 (Extremely Satisfied). Total score ranges from 1 to 7. Higher score indicate improvement.
Time Frame: Baseline and endpoint Part 2 (up to 9 Months)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part-2: Paliperidone Palmitate (PP) | Part-2: OAP
Number analyzed (Participants) | 73 | 156
units on a scale | -0.2 (1.44) | 0.1 (1.16)

17. Secondary Outcome: Part 3 (EDP): Change From Baseline in Functioning as Measured by the Personal and Social Performance (PSP) Total Score
Description: as for outcome 5
Time Frame: Baseline and 18 Months
Population: Analysis was performed on part 3 ITT analysis set. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Part 3-PP to PP | Part 3-OAP to OAP
Number analyzed (Participants) | 41 | 47
units on a scale | 7.5 (1.94) | 7.0 (1.82)

18. Secondary Outcome: Part 3 (EDP): Change From Baseline in Adjusted Intracortical Myelin Fraction Score as Measured by Inversion Recovery (IR) and Spin Echo Magnetic Resonance Imaging (MRI)
Description: as for outcome 6
Time Frame: Baseline and 18 Months
Population: Analysis was performed on Part 3 ITT analysis set.
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Part 3-PP to PP | Part 3-OAP to OAP
Number analyzed (Participants) | 49 | 63
ratio | -0.001 (0.001) | -0.003 (0.001)

19. Secondary Outcome: Part 3 (EDP): Time to First Treatment Failure
Description: as for outcome 1
Time Frame: From Day 1 Up to 18 Months
Population: Analysis was performed on Part 3 ITT analysis set.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part 3-PP to PP | Part 3-OAP to OAP
Number analyzed (Participants) | 49 | 63
days | NA [NA to NA] — Here, NA signifies that median and upper/lower limit of CI was not estimable due to less number of events. | NA [376.0 to NA] — Here, NA signifies that median and upper/lower limit of CI was not estimable due to less number of events.

20. Secondary Outcome: Part 3 (EDP): Change From Baseline in Working Memory Score: MCCB Domain
Description: as for outcome 7
Time Frame: Baseline and 18 Months
Population: Analysis was performed on Part 3 ITT analysis set.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Part 3-PP to PP | Part 3-OAP to OAP
Number analyzed (Participants) | 49 | 63
T-score | -1.7 (1.24) | 0.7 (1.16)

21. Secondary Outcome: Part 3 (EDP): Change From Baseline in Verbal Learning Score: MCCB Domain
Description: as for outcome 8
Time Frame: Baseline and 18 Months
Population: Analysis was performed on Part 3 ITT analysis set.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Part 3-PP to PP | Part 3-OAP to OAP
Number analyzed (Participants) | 49 | 63
T-score | 0.3 (1.24) | 0.8 (1.15)

22. Secondary Outcome: Part 3 (EDP): Change From Baseline in Speed of Processing Score: MCCB Domain
Description: MCCB measures cognitive function across cognitive domains and is comprised of 10 independent tests assessing 7 cognitive domains (speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition). A subset of the MCCB cognitive domain was used to assess speed of processing score of participants. The range of speed of processing score T-scores for a normal control population is between 0 to 100 with a mean of 50 and standard deviation of 10. Higher scores indicate better cognitive functioning.
Time Frame: Baseline and 18 Months
Population: Analysis was performed on Part 3 ITT analysis set.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Part 3-PP to PP | Part 3-OAP to OAP
Number analyzed (Participants) | 49 | 63
T-score | 2.5 (1.32) | 4.9 (1.24)

23. Secondary Outcome: Part 3 (EDP): Change From Baseline in Attention/Vigilance Score: MCCB Domain
Description: as for outcome 10
Time Frame: Baseline and 18 Months
Population: Analysis was performed on Part 3 ITT analysis set.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Part 3-PP to PP | Part 3-OAP to OAP
Number analyzed (Participants) | 49 | 63
T-score | 2.4 (1.46) | 0.7 (1.35)

24. Secondary Outcome: Part 3 (EDP): Change From Baseline in Visual Learning Score: MCCB Domain
Description: as for outcome 11
Time Frame: Baseline and 18 Months
Population: Analysis was performed on Part 3 ITT analysis set.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Part 3-PP to PP | Part 3-OAP to OAP
Number analyzed (Participants) | 49 | 63
T-score | 0.2 (1.42) | -0.2 (1.35)

25. Secondary Outcome: Part 3 (EDP): Change From Baseline in Reasoning and Problem Solving: MCCB Domain
Description: MCCB measures cognitive function across cognitive domains and is comprised of 10 independent tests assessing 7 cognitive domains (speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition). A subset of the MCCB cognitive domain was used to assess reasoning and problem solving score of participants. The range of reasoning and problem solving T-scores for a normal control population is between 0 to 100 with a mean of 50 and standard deviation of 10. Higher scores indicate better cognitive functioning.
Time Frame: Baseline and 18 Months
Population: Analysis was performed on Part 3 ITT analysis set.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Part 3-PP to PP | Part 3-OAP to OAP
Number analyzed (Participants) | 49 | 63
T-score | 3.4 (1.46) | 4.7 (1.34)

26. Secondary Outcome: Part 3 (EDP): Change From Baseline in Social Cognition Score: MCCB Domain
Description: as for outcome 13
Time Frame: Baseline and 18 Months
Population: Analysis was performed on Part 3 ITT analysis set.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Part 3-PP to PP | Part 3-OAP to OAP
Number analyzed (Participants) | 49 | 63
T-score | -0.2 (1.36) | 1.4 (1.26)

27. Secondary Outcome: Part 3 (EDP): Change From Baseline in Clinical Global Impression Severity (CGI-S) Score
Description: The Clinical Global Impression Severity (CGI-S) rating scale is used to rate the severity of a participant's overall clinical condition on a 7 point scale. The total score ranges from 1 to 7, where 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill participants". Higher scores indicate worsening.
Time Frame: Baseline, up to 18 Months
Population: Analysis was performed on Part 3 ITT analysis set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part 3-PP to PP | Part 3-OAP to OAP
Number analyzed (Participants) | 49 | 63
units on a scale | -0.7 (0.14) | -0.7 (0.14)

28. Secondary Outcome: Part 3 (EDP): Number of Participants With Change From Baseline in Severity of Psychotic Symptoms, as Measured by CRDPSS
Description: as for outcome 15
Time Frame: Baseline, up to 18 Months
Population: Analysis was performed on Part 3 ITT analysis set. Here, N (number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3-PP to PP | Part 3-OAP to OAP
Number analyzed (Participants) | 41 | 47
Participants
  Hallucinations: Worsened | 3 | 8
  Hallucinations: Unchanged | 27 | 29
  Hallucinations: Improved | 11 | 10
  Delusions: Worsened | 6 | 10
  Delusions: Unchanged | 21 | 20
  Delusions: Improved | 14 | 17
  Disorganized Speech: Worsened | 2 | 3
  Disorganized Speech: Unchanged | 27 | 36
  Disorganized Speech: Improved | 12 | 8
  Abnormal Psychomotor Behavior: Worsened | 4 | 2
  Abnormal Psychomotor Behavior: Unchanged | 32 | 37
  Abnormal Psychomotor Behavior: Improved | 5 | 8
  Negative Symptoms: Worsened | 11 | 4
  Negative Symptoms: Unchanged | 11 | 22
  Negative Symptoms: Improved | 19 | 21
  Impaired Cognition: Worsened | 10 | 9
  Impaired Cognition: Unchanged | 14 | 23
  Impaired Cognition: Improved | 17 | 15
  Mania: Worsened | 0 | 3
  Mania: Unchanged | 40 | 39
  Mania: Improved | 1 | 5
  Depression: Worsened | 7 | 6
  Depression: Unchanged | 26 | 29
  Depression: Improved | 8 | 12

29. Secondary Outcome: Part 3 (EDP): Change From Baseline in Medication Satisfaction Questionnaire (MSQ) Score
Description: as for outcome 16
Time Frame: Baseline, up to 18 Months
Population: Analysis was performed on part 3 ITT analysis set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part 3-PP to PP | Part 3-OAP to OAP
Number analyzed (Participants) | 49 | 63
units on a scale | 0.3 (0.18) | 0.4 (0.18)

30. Secondary Outcome: Part 3 (Disease Modification): Personal and Social Performance (PSP) Total Observed Score
Description: The Personal and Social Performance (PSP) scale assesses degree of a participant's dysfunction within 4 domains of behavior: 1) socially useful activities, 2) personal and social relationships, 3) self-care, and 4) disturbing and aggressive behavior. Score ranges from 1 to 100, divided into 10 equal intervals to rate degree of difficulty (1 = absent, 2 = mild, 3 = manifest, 4 = marked, 5 = severe, and 6 = very severe) in each of the 4 domains. Based on 4 domains there will be 1 transformed total score. Participants with score of 71 to 100 have mild degree of difficulty; from 31 to 70, varying degrees of disability; less than or equal to 30, functioning so poorly as to require intensive supervision.
Time Frame: Month 9 of Part 3
Population: Analysis was performed on Part 3 ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Part 3-PP to PP | Part 3- OAP to PP (or Delayed-Start PP) | Part 3-OAP to OAP
Number analyzed (Participants) | 49 | 57 | 63
units on a scale | 67.6 (1.81) | 66.1 (1.70) | 66.6 (1.70)

31. Secondary Outcome: Part 3 (Disease Modification): Change From Baseline in Adjusted Intracortical Myelin Fraction Score as Measured by Inversion Recovery (IR) and Spin Echo Magnetic Resonance Imaging (SE MRI)
Description: as for outcome 6
Time Frame: Baseline and Month 9 of Part 3
Population: Analysis was performed on Part 3 ITT analysis set. Here 'N' (number of participants analyzed) signifies number of participants analyzed for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Part 3-PP to PP | Part 3- OAP to PP (or Delayed-Start PP) | Part 3-OAP to OAP
Number analyzed (Participants) | 10 | 8 | 9
ratio | -0.7 (1.02) | -0.2 (0.95) | 0.5 (0.96)

ADVERSE EVENTS:
Time Frame: Up to 20 Months
Description: Safety analysis was based on Part 1, 2 and 3 Intent-to-Treat (ITT) analysis set. Part 1, 2 and 3 ITT analysis set included all randomized subjects who received at least one dose of study medication (or any portion of the dose) in Part 1, 2 and 3 regardless of their compliance with the protocol.
Arm/Group | Part 1-Run-in: Oral Antipsychotics (OAP) | Part 2-Paliperidone Palmitate (PP) | Part 2-OAP | Part 3-PP to PP (Extended Disease Progression [EDP] and Disease Modification) | Part 3- OAP to PP (or Delayed-Start PP) (Disease Modification) | Part 3-OAP to OAP (EDP and Disease Modification)
All-Cause Mortality (participants affected / at risk) | 0/273 | 1/78 | 0/157 | 0/49 | 0/57 | 0/63
Serious Adverse Events (participants affected / at risk) | 10/273 | 10/78 | 19/157 | 1/49 | 3/57 | 8/63
Other Adverse Events (participants affected / at risk) | 116/273 | 50/78 | 89/157 | 18/49 | 34/57 | 27/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1-Run-in: Oral Antipsychotics (OAP) (N=273) | Part 2-Paliperidone Palmitate (PP) (N=78) | Part 2-OAP (N=157) | Part 3-PP to PP (Extended Disease Progression [EDP] and Disease Modification) (N=49) | Part 3- OAP to PP (or Delayed-Start PP) (Disease Modification) (N=57) | Part 3-OAP to OAP (EDP and Disease Modification) (N=63)
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Exposure Via Inhalation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0
Ganglioglioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Catatonia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Completed Suicide (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Depressed Mood (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Homicidal Ideation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Mania (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mental Status Changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Psychotic Disorder (Psychiatric disorders) | 1 | 4 | 5 | 0 | 0 | 4
Psychotic Symptom (Psychiatric disorders) | 1 | 0 | 3 | 0 | 0 | 2
Schizophrenia (Psychiatric disorders) | 3 | 3 | 6 | 0 | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 0 | 3 | 4 | 0 | 2 | 0
Suicide Attempt (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1-Run-in: Oral Antipsychotics (OAP) (N=273) | Part 2-Paliperidone Palmitate (PP) (N=78) | Part 2-OAP (N=157) | Part 3-PP to PP (Extended Disease Progression [EDP] and Disease Modification) (N=49) | Part 3- OAP to PP (or Delayed-Start PP) (Disease Modification) (N=57) | Part 3-OAP to OAP (EDP and Disease Modification) (N=63)
Nausea (Gastrointestinal disorders) | 5 | 4 | 11 | 2 | 2 | 5
Fatigue (General disorders) | 10 | 4 | 1 | 0 | 5 | 1
Injection Site Pain (General disorders) | 4 | 6 | 2 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 5 | 4 | 3 | 0 | 4
Upper Respiratory Tract Infection (Infections and infestations) | 6 | 1 | 7 | 1 | 3 | 2
Blood Prolactin Increased (Investigations) | 8 | 3 | 9 | 1 | 0 | 1
Weight Increased (Investigations) | 44 | 22 | 50 | 7 | 9 | 5
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 2 | 4 | 3 | 0 | 1 | 2
Akathisia (Nervous system disorders) | 10 | 7 | 8 | 0 | 4 | 0
Headache (Nervous system disorders) | 11 | 7 | 12 | 1 | 2 | 4
Sedation (Nervous system disorders) | 16 | 3 | 3 | 0 | 2 | 0
Somnolence (Nervous system disorders) | 19 | 7 | 4 | 1 | 3 | 1
Tremor (Nervous system disorders) | 6 | 1 | 7 | 2 | 5 | 2
Anxiety (Psychiatric disorders) | 5 | 5 | 4 | 0 | 6 | 3
Insomnia (Psychiatric disorders) | 9 | 4 | 9 | 5 | 6 | 4
Paranoia (Psychiatric disorders) | 0 | 0 | 0 | 3 | 0 | 1
Schizophrenia (Psychiatric disorders) | 3 | 1 | 4 | 1 | 3 | 1

LIMITATIONS AND CAVEATS:
The treatment failure (TF) definition for this study was very broad. For example, the TF reason, supplementation with another antipsychotic, was biased against PP as supplementing with oral paliperidone or risperidone was considered a TF which is usual clinical practice. Supplementation was the most common first TF criteria for PP. A designated individual of the subject was a requirement for study inclusion which may have also contributed to increased OAP adherence in the beginning of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-11-02): https://cdn.clinicaltrials.gov/large-docs/02/NCT02431702/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-06): https://cdn.clinicaltrials.gov/large-docs/02/NCT02431702/SAP_001.pdf